CLINICAL TRIAL: NCT07271784
Title: Establishment of a Prediction Model for Postherpetic Neuralgia Based on Immune Cell Typing
Brief Title: Establishment of a Prediction Model for Postherpetic Neuralgia
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhiying Feng, Director of the Pain Department, First Affiliated Hospital of Zhejiang University
Other Study IDs: [2023B] IIT.No.0673
Record Dates: First submitted 2025-09-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pain; Neuropathic Pain; Biomarkers / Blood
Keywords: Postherpetic neuralgia; biomarker
MeSH Terms: conditions — Pain; Neuralgia; Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHN Group: Patients with herpes zoster were classified into the postherpetic neuralgia (PHN) group if they had a Numerical Rating Scale (NRS) pain score ≥1 at 3 months after disease onset.
- non-PHN Group: Patients with herpes zoster were classified into the non postherpetic neuralgia (non-PHN) group if they had a Numerical Rating Scale (NRS) pain score of 0 at 3 months after disease onset.

SUMMARY:
This prospective cohort study enrolled 300 herpes zoster (HZ) patients at varying disease stages (1 week to 3 months post-onset) to investigate predictors of postherpetic neuralgia (PHN). Comprehensive baseline data were collected, including demographic characteristics (age, sex, body mass index [BMI]), clinical comorbidities (hypertension, diabetes mellitus), disease-specific parameters (duration of zoster-associated pain [ZAP], dermatomal distribution, pregabalin dosage equivalents), and psychometric assessments using validated scales (Numerical Rating Scale [NRS], age-adjusted Charlson Comorbidity Index [aCCI], Generalized Anxiety Disorder-7 [GAD-7], Patient Health Questionnaire-9 [PHQ-9], and Insomnia Severity Index [ISI]). Laboratory evaluations encompassed routine hematological tests (complete blood count [CBC], hepatic/renal function), metabolic profiling (triglycerides [TG], total cholesterol [TC], lipoprotein subfractions), inflammatory markers (erythrocyte sedimentation rate [ESR], comprehensive cytokine panel including interleukins [IL] and interferons [IFN]), and detailed immunophenotyping via multicolor flow cytometry of peripheral blood lymphocytes. After a 3-month follow-up, patients were to be stratified into PHN and non-PHN groups based on pain persistence. The use of least absolute shrinkage and selection operator (LASSO) regression analysis was planned to identify significant predictive factors and develop a multivariate model, with the aim of establishing a precision medicine framework for early PHN risk stratification through integrated analysis of clinical and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years Location of pain consistent with the HZ region and pain originating from herpes zoster (HZ)

Exclusion Criteria:

Mental disorders, cognitive deficits, or coexisting painful diseases Severe cardio-cerebrovascular disease, hepatorenal insufficiency, infectious disease Cancer with a recurrence-free survival of less than one year Hematological disorders such as lymphoma or conditions such as acquired immune deficiency syndrome (AIDS) Psychiatric disorders; alcohol addiction; opioid abuse Previous treatment with interventional neurodestructive therapies or spinal cord stimulation (SCS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects included patients with zoster associated pain who meet the inclusion and exclusion criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of Postherpetic Neuralgia (PHN) as Assessed by the Numerical Rating Scale (NRS) at 3 months after herpes zoster onset. | At the 3-month timepoint after herpes zoster onset.
  HN is defined as pain that persists in the area affected by the herpes zoster rash after the acute rash has healed, and that is present at 3 months after rash onset. The presence and intensity of this pain will be assessed using the Numerical Rating Scale (NRS), with an NRS score of ≥ 1 used as the threshold to define the presence of clinically pain. Study participants will be categorized based on the presence of PHN at the 3-month timepoint according to this definition.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No